CLINICAL TRIAL: NCT07245342
Title: Early Electroacupuncture for Urinary Continence After Radical Prostatectomy: A Randomized, Single-Blind, Sham-Electroacupuncture-Controlled, Parallel-Group, Multicenter Clinical Trial
Brief Title: Electroacupuncture for Improving Urinary Incontinence After Radical Prostatectomy
Acronym: EA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiangyang Zhan, Physician in Charge, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-1593-176-01
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Electroacupuncture; Prostate Cancer; Radical Prostatectomy; Urinary Continence Recovery
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture Group (Experimental): Patients in this group will receive electroacupuncture intervention starting from 1 week after radical prostatectomy, following a standardized treatment schedule to assess its effect on postoperative urinary continence recovery.
  Interventions: Procedure: Electroacupuncture
- Sham Electroacupuncture Group (Placebo Comparator): Patients in this group will receive sham electroacupuncture intervention with the same treatment schedule and duration as the electroacupuncture group, to serve as a placebo control and ensure the validity of the trial results.
  Interventions: Procedure: Sham Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Bilateral acupoints Shangliao (BL31), Ciliao (BL32), Zhongliao (BL33), Xialiao (BL34), and Shenshu (BL23) were localized according to WHO standards. Following skin disinfection, each point was punctured using a sterile disposable needle (0.30 × 45 mm) and manually stimulated via lifting, thrusting, and rotating for 30 seconds to elicit deqi. An electroacupuncture device (SDZ-II, Huatuo brand) was then connected, delivering continuous wave stimulation at 50 Hz. Current intensity was set between 1-5 mA to produce mild local muscle trembling without pain, applied for 20 minutes per session.Treatments were administered three times weekly (preferably every other day) for six weeks. All procedures were performed by licensed acupuncturists with ≥2 years of experience, who received standardized pre-trial training in point localization, needling technique, and device operation.
  Arms: Electroacupuncture Group
Procedure: Sham Electroacupuncture — Patients in the control group will receive sham acupuncture identical in schedule and duration to the electroacupuncture group. Needling will be performed at non-acupoint sites, 1 cun lateral to the true acupoints (BL31-BL34, BL23), using superficial insertion (1-4 mm depth) without manual stimulation to prevent deqi.A deactivated electroacupuncture device (SDZ-II, Huatuo brand) with internally short-circuited wiring will be attached to mimic the active treatment setup, though no current will be delivered.All sham acupuncture procedures will be conducted by licensed acupuncturists with at least two years of experience, who will receive standardized training prior to the trial in sham point location and needling protocols to ensure procedural consistency.
  Arms: Sham Electroacupuncture Group

SUMMARY:
This clinical trial aims to find out if early electroacupuncture (EA) helps people recover the ability to control urination and is safe after surgery to remove the prostate gland for prostate cancer (radical prostatectomy).

Participants are people aged 18 to 80 with localized prostate cancer who have had radical prostatectomy and are in good physical condition (ECOG score 0-1, meaning they can manage daily activities well).

It will answer two key questions:

Does early EA make more people fully control their urination 3 months after prostate surgery? How does early EA affect urination control and safety at 1, 6, and 12 months after surgery? Researchers will compare two groups: one getting EA and the other getting a fake version (sham EA ) to see if EA works better.

Participants will start treatment 1 week after surgery, getting EA or sham EA 3 times a week for 6 weeks, 20 minutes each time. They will also complete tests to check urination control and fill out surveys about their urination, quality of life, and symptoms at different times. Their safety will be watched closely too.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most commonly diagnosed malignancy and the second leading cause of cancer-related death among men worldwide, significantly impacting both physical and psychological health. Radical prostatectomy (RP) remains the gold standard for treating localized prostate cancer, with three primary goals: oncologic control, recovery of urinary continence, and preservation of sexual function. While advances in surgical techniques and pharmacotherapy have substantially improved cancer control outcomes, functional recovery-particularly regarding post-prostatectomy incontinence (PPI)-remains a major challenge. PPI primarily results from intraoperative damage to the bladder neck structure and surrounding nerves, compromising urinary control. Postoperative ischemia and scar adhesion may further exacerbate incontinence. Studies report PPI rates of 18%-55% at 3 months and 4%-31% at 1 year after RP. Electroacupuncture(EA), evolved from traditional manual acupuncture, augments the technique by applying controlled electrical currents. Evidence suggests that EA can deliver pulsed currents to stimulate muscles and nerves, inducing passive contractions of the pelvic floor muscles. It may also excite sympathetic nerves, inhibit parasympathetic activity, modulate detrusor contractility, enhance urethral sphincter function, and improve urethral closure-all of which may contribute to restoring urinary control.Given these potential benefits, along with its simplicity, low cost, and favorable safety profile, we hypothesize that early post-surgical EA-initiated immediately after RP-may promote urinary continence more effectively than delayed intervention after conservative treatments have failed. This approach aligns with both clinical needs and the traditional Chinese medicine principle of "preventive treatment."Based on the premise that early EA can accelerate the recovery of urinary continence after RP, we previously conducted an observational study. The results indicated that early EA was associated with higher rates of early complete continence recovery, shorter time to continence, and high patient satisfaction, with no reported adverse events.To further evaluate the efficacy and safety of early EA for PPI, we designed this randomized, single-blind, sham-controlled, multicenter trial. Patients undergoing robotic or laparoscopic RP will be assigned to either EA or sham EA, with intervention starting within one week post-surgery and lasting for six weeks. The study aims to assess efficacy and safety outcomes, thereby determining whether early EA facilitates urinary continence recovery in patients following RP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years (inclusive) with a diagnosis of localized prostate cancer scheduled for radical prostatectomy.
2. Clinical tumor stage ≤ cT2bN0M0 confirmed by preoperative evaluation.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Willingness to participate in the study and provision of written informed consent.

Exclusion Criteria:

1. Presence of preoperative detrusor overactivity, urethral stricture, urge urinary incontinence, stress urinary incontinence, or overflow urinary incontinence.
2. Preoperative International Prostate Symptom Score (IPSS) ≥ 20.
3. Concurrent urogenital infectious diseases (e.g., acute urethritis, acute cystitis).
4. History of pelvic radiotherapy.
5. Previous prostate surgery.
6. Severe cardiovascular disease, hepatic or renal dysfunction, or coagulation disorders.
7. Presence of psychiatric or psychological conditions impairing the ability to provide coherent feedback.
8. Receipt of any acupuncture treatment within one month prior to the study.
9. Needle phobia, history of fainting during acupuncture, or strong aversion to acupuncture therapy.
10. Any other condition considered by the investigators to render the patient unsuitable for study participation.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2028-11-25 (Estimated); Study Completion 2029-02-25 (Estimated)

PRIMARY OUTCOMES:
Complete Urinary Continence Rate | 3 months postoperatively
  The proportion of patients achieving complete urinary continence (defined as ≤1 safety pad per day).

SECONDARY OUTCOMES:
Complete Urinary Continence Rate | 1, 6, and 12 months postoperatively
  The proportion of patients achieving complete urinary continence (defined as ≤1 safety pad per day).
International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI-SF) score | 1, 3, 6, and 12 months postoperatively
  The International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI-SF) is used to assess the impact of urinary incontinence on quality of life over the past four weeks. It comprises three scored items addressing the frequency of leakage, the amount of leakage, and the overall impact on daily life, along with a fourth unscored item designed to help determine the type of incontinence. The total score ranges from 0 to 21, with higher scores indicating greater severity.
Incontinence-Quality of Life (I-QOL) Questionnaire score | 1, 3, 6, and 12 months postoperatively
  Scores are inversely related to symptom severity, meaning a higher score denotes a superior quality of life.
Visual Analog Scale (VAS) | 1, 3, 6, and 12 months postoperatively
  Scored by measuring the patient's mark on a 10-cm line, where a greater length indicates poorer self-rated urinary control.
King's Health Questionnaire (KHQ) score | 1, 3, 6, and 12 months postoperatively
  The King's Health Questionnaire (KHQ) is a condition-specific instrument for assessing quality of life in individuals with urinary incontinence. It evaluates multiple domains, including role, physical, and social limitations, personal relationships, emotions, and symptom severity.
International Prostate Symptom Score (IPSS) | 1, 3, 6, and 12 months postoperatively
  The International Prostate Symptom Score (IPSS) is a patient-reported instrument that assesses the severity of lower urinary tract symptoms (LUTS). The total score ranges from 0 to 35, with categories defined as mild (0-7), moderate (8-19), and severe (20-35).
Quality of Life Core Questionnaire (QLQ-C30) score | 1, 3, 6, and 12 months postoperatively
  The EORTC QLQ-C30 is a validated, cancer-specific instrument for assessing health-related quality of life. It comprises 30 items across several functional scales, symptom scales, and a global health status scale.
Analysis of Risk Factors Influencing Treatment Efficacy (Multivariable Logistic Regression) | 3 months postoperatively
  Through multivariate logistic regression analysis, evaluate the impact of factors such as age, BMI, underlying diseases, and surgical methods on the efficacy of early EA treatment for urinary incontinence (cured or not).
Median Time to Complete Urinary Continence | Within 12 months postoperatively
  Time from radical prostatectomy to the first day of maintaining complete urinary continence (defined as using 0 or 1 pad per day), assessed at follow - up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyang Zhan, Principal Investigator — Shuguang Hospital Affiliated to Shanghai University of Chinese Medicine

IPD SHARING:
Plan to Share IPD: No